CLINICAL TRIAL: NCT05999890
Title: A Comparative Study Between Intranasal Tapentadol Versus Intravenous Paracetamol for Post-operative Analgesia in Lower Limb Orthopedic Surgeries Under Spinal Anaesthesia'
Brief Title: Comparison of Postoperative Analgesia Between Intravenous Paracetamol and Intranasal Tapentadol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kempegowda Institute of Medical Sciences, Bangalore (Other Government)
Responsible Party: Principal Investigator, Priyanka Suresh, Assistant Professor, Kempegowda Institute of Medical Sciences, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KIMS/IEC/A035/D/2021; NCT05967221 (obsolete NCT alias)
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Lower Limb Fracture
MeSH Terms: interventions — Tapentadol; Acetaminophen

STUDY DESIGN:
Intervention Model Description: It is a single blind randomized controlled trial comparing the intranasal tapentadol with intravenous paracetamol for post operative analgesia
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor) The assessor of the outcome would measure hemodynamic parameters and severity of the pain at the mentioned time intervals. The assessor was not involved in the randomization / administration of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tapentadol (Experimental): Tapentadol is a novel, centrally acting analgesic with dual mechanism of action, combining mu-opioid receptor agonism with norepinephrine reuptake inhibition.this dual mode of action is responsible for its opioid sparing effect, which contributes to reduction in some of the typical opioid related adverse effects
  Interventions: Drug: Tapentadol Hydrochloride
- Paracetamol (Active Comparator): Paracetamol is one of the most frequently used analgesic and antipyretic agent, interferes neither with platelet nor kidney functions nor does it present the unwanted side effects of NSAIDS.
  Interventions: Drug: Tapentadol Hydrochloride

INTERVENTIONS:
Drug: Tapentadol Hydrochloride — Intranasal administration of tapentadol was compared with intravenous paracetamol for postoperative analgesia
  Other Names: Paracetamol

SUMMARY:
The aim of the study was to compare the analgesic efficacy of intranasal tapentadol nasal spray 44.5mg and intravenous paracetamol 1gm during the postoperative period by Visual analog scale(VAS)in patients undergoing lower limb(long bone fractures)orthopedic surgeries. Paracetamol is one of the most frequently used analgesic and antipyretic agents, interferes neither with platelet nor kidney functions nor does it present the unwanted side effects of NSAIDs. Tapentadol is a novel, centrally-acting analgesic with a dual mechanism of action, combining mu-opioid receptor agonism with norepinephrine reuptake inhibition. This dual mode of action is responsible for its opioid-sparing effect, which contributes to a reduction in some of the typical opioid-related adverse effects

DETAILED DESCRIPTION:
Inclusion criteria Age: From 18.00 Year(s) to 60.00 years Gender: Both American Society of Anesthesiologists (ASA) physical status: 1 & 2, posted for elective lower limb orthopedic surgeries Exclusion criteria

1. Sepsis at the site of injection
2. Coagulopathy
3. Patients with history of renal, hepatic, cardiovascular disease
4. Patient on chronic opioid use Outcome Comparing postoperative analgesia between the groups every 12 hours after the intervention till about 72 hours post intervention. The secondary outcome is to compare the need for the rescue analgesia between the groups

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status 1 & 2
2. Posted for elective lower limb orthopaedic surgeries

Exclusion Criteria:

1. Sepsis at the site of injection
2. Coagulopathy
3. Patients with history of renal, hepatic, cardiovascular disease
4. Patient on chronic opioid use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Pain as measured with Visual analogue scale | Every 12 hours after the intervention till about 72 hours after the intervention
  The pain rating was done as per a visual analogue scale (VAS) of 0-100 (score 0 = no pain, score 100 - most severe pain). Patients with a VAS score of more than 30, at what is considered as base line, in group A=received IV paracetamol 1gm given every 5-6 hourly and in group B=received intranasal tapentadol 44.5mg nasal spray administered every 5-6 hourly. Patient was assessed for pain by using VAS half an hour after administration and the scores were documented. Pain score were recorded at and after 30 minutes of the intervention in the following time frames - 12hr,24hr,36hr,48hr, 60hr and 72hrs after the baseline intervention (0hr).

SECONDARY OUTCOMES:
The need for rescue analgesia | In the first 72 hours after the initiation of the intervention
  The need for the add on analgesic whenever the subjects request for the same

CONTACTS AND LOCATIONS:
Locations (1):
- Kempegowda Institute of Medical Sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared; If needed only anonymised individual data will be shared